CLINICAL TRIAL: NCT00792181
Title: Intervention Study to Relieve Pain and Anxiety in Acute Myocardial Disease Focusing on Treatment With Benzodiazepines(Midazolam)and the Importance of a Caring Relation.
Brief Title: To Relieve Pain and Anxiety - an Intervention Study in Ambulance Services
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Med. doctor, Medical Products Agency - Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPA Dnr 151:2008/4564
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2008-11-17 (Estimated); Status verified 2008-11

CONDITIONS: Acute Myocardial Infarction; Pain
Keywords: The focus is the pain reduce in the first 15 minutes for patients suffering an acute myocardial infarction, treated by caregivers in Ambulance service.
MeSH Terms: conditions — Pain | interventions — Midazolam; Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Medical intervention - with benzodiazepines (Midazolam).
  Interventions: Drug: Midazolam
- 2 (Experimental): Course intervention - a professional development course for caregivers.
  Interventions: Other: Course intervention - a professional development course for caregivers.
- 3 (Experimental): Combination of both medical interventions and a professional development course for caregivers.
  Interventions: Drug: Midazolam; Other: Course intervention - a professional development course for caregivers.
- 4 (No Intervention): No intervention at all = a control group

INTERVENTIONS:
Drug: Midazolam — Midazolam 1 mg: 70 years or more and less than 70 kg Midazolam 2 mg: under 70 years and 70 kg or more
  Arms: 1; 3
Other: Course intervention - a professional development course for caregivers. — The nursing intervention involves a professional development course for caregivers. The course is expected to deepen the caregivers' knowledge about the encounter with patients as well as cardiovascular treatment.
  Arms: 2; 3

SUMMARY:
This is an intervention study focusing on both medical and nursing questions. The study is a joint project between the Ambulance services at four cities in West Sweden and Knowledge and research centre, PreHospen at University of Borås. The aim is to prove the importance of a caring relation between a patient and a caregiver in cases when a caregiver treats a patient with benzodiazepines (Midazolam). The overall aim is to show that knowledge and skills in both caring science and medicine can be applied at the same time in order to relieve pain and anxiety in acute myocardial disease.

The nursing intervention involves a professional development course for caregivers. The course is expected to deepen the caregivers' knowledge about the encounter with patients as well as cardiovascular treatment.

Following questions are formulated:

A. What are the effects regarding relieving pain and anxiety in acute myocardial disease? B. What are the effects regarding circulatory influence? C. What are the effects regarding patients' experiences of the ambulance services? D. What are the effects regarding number of care days in relation to acute myocardial disease? E. What are the effects of patients' disease complications?

ELIGIBILITY:
Inclusion Criteria:

1. Patients in Ambulance service with chest pain and suspicion about acute coronary syndrome.
2. At least 4 on a Coloured Analogue Scale.

Exclusion Criteria:

1. Blood pressure less than 100 mmHg
2. Children under 18 years
3. Under the influence of alcohol
4. Under the influence of drugs
5. Treatment with benzodiazepines
6. Disorientated
7. Communication problems
8. Trauma

Age Groups: Child, Adult, Older Adult
Enrollment: 2800 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual)

REFERENCES:
- [Derived] Holmberg M, Andersson H, Winge K, Lundberg C, Karlsson T, Herlitz J, Wireklint Sundstrom B. Association between the reported intensity of an acute symptom at first prehospital assessment and the subsequent outcome: a study on patients with acute chest pain and presumed acute coronary syndrome. BMC Cardiovasc Disord. 2018 Nov 28;18(1):216. doi: 10.1186/s12872-018-0957-3. PMID 30486789
- [Derived] Wireklint Sundstrom B, Holmberg M, Herlitz J, Karlsson T, Andersson H. Possible effects of a course in cardiovascular nursing on prehospital care of patients experiencing suspected acute coronary syndrome: a cluster randomised controlled trial. BMC Nurs. 2016 Sep 2;15(1):52. doi: 10.1186/s12912-016-0175-1. eCollection 2016. PMID 27594805